CLINICAL TRIAL: NCT03088605
Title: A Single-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of TOP1630 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye Syndrome
Brief Title: Safety and Efficacy of TOP1630 for Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Collaborators: Topivert Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOP1630-TV-04
Record Dates: First submitted 2017-03-10; First posted 2017-03-23 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): TOP1630 Ophthalmic Solution
  Interventions: Drug: TOP1630 Ophthalmic Solution
- Placebo (Placebo Comparator): Placebo (Vehicle) Ophthalmic Solution
  Interventions: Drug: Placebo to TOP1630 Ophthalmic Solution

INTERVENTIONS:
Drug: TOP1630 Ophthalmic Solution — Bilateral ocular drug administration
  Arms: Active
Drug: Placebo to TOP1630 Ophthalmic Solution — Bilateral ocular drug administration
  Arms: Placebo

SUMMARY:
In subjects with Dry Eye Syndrome:

The primary objective of this study is to compare the safety and tolerability of TOP1630 Ophthalmic Solution to placebo.

The secondary objectives are to compare the efficacy of TOP1630 Ophthalmic Solution to placebo for the treatment of the signs and symptoms of dry eye syndrome.

DETAILED DESCRIPTION:
This study is designed to assess the safety, tolerability and efficacy of TOP1630 ophthalmic solution in subjects with Dry Eye Syndrome.

Eligible subjects will be randomized double masked to either TOP1630 or placebo.

Part 1 (time frame 12 days) comprises assessment of safety, tolerability and ocular comfort.

Part 2 (time frame 35 days) comprises assessment of safety, tolerability and efficacy

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a reported history of dry eye;
* Have a history of use of eye drops for dry eye symptoms;

Additionally for Part 2

Symptoms of dry eye syndrome including:

* Ocular discomfort
* Conjunctival redness
* Tear film break up time
* Schirmer test score

Signs of dry eye syndrome including:

Conjunctival staining score

Exclusion Criteria:

* Have any clinically significant slit lamp findings at entry visit ;
* Be diagnosed with an ongoing ocular infection;
* Have any significant ocular lesion that could interfere with assessment of safety or efficacy or prevent study conduct in the opinion of the PI;
* Have any planned ocular and/or lid surgeries over the study period;
* Have an uncontrolled systemic disease;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;
* Have a known allergy and/or sensitivity to the test article or its components;
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Placebo
Started | 37 | 32
Completed | 36 | 32
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.42) | 65.3 (11.92) | 63.9 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 11 | 14 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 28 | 59
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual Acuity will be measured using the EDTRS chart to assess changes from baseline
Time Frame: Part 1: 12 days time frame; Part 2: 35 days time frame
Population: Number analyzed represents the sum of numbers analyzed Part 1 and Part 2
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Active | Placebo
Number analyzed (Participants) | 37 | 32
logMAR
  Part 1: number analyzed (Participants) | 6 | 2
  Part 1 | 0.05 (0.143) | -0.09 (0.156)
  Part 2: number analyzed (Participants) | 31 | 30
  Part 2 | 0.017 (0.1163) | 0.075 (0.1242)

2. Primary Outcome: Slit-lamp Biomicroscopy
Description: Slit lamp biomicroscopy exams will be performed to assess any changes from baseline; outcome measure is number of patients with no abnormalities
Time Frame: Part 1: 12 days time frame; Part 2: 35 days time frame
Measure: Number; unit: participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 37 | 32
participants
  Part 1 | 6 | 2
  Part 2 | 31 | 30

3. Primary Outcome: Drop Comfort Assessment
Description: The comfort of the eye drop will be performed to assess changes from baseline. Drop Comfort Assessment Scale; 0-10; 0 being very comfortable and 10 being very uncomfortable
Time Frame: Part 1: 12 days time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 6 | 2
score on a scale | 0.71 (0.846) | 1.38 (0.495)

4. Primary Outcome: Intraocular Pressure
Description: a non-contact tonometer will be used to perform IOP to assess changes from baseline.
Time Frame: Part 1: 12 days time frame; Part 2: 35 days time frame
Population: Number analyzed comes from Part 1 and Part 2
Measure: Mean (Standard Deviation); unit: unit of measure "mmHg"
Arm/Group | Active | Placebo
Number analyzed (Participants) | 37 | 32
unit of measure "mmHg"
  Part 1: number analyzed (Participants) | 6 | 2
  Part 1 | 12.3 (1.03) | 15.5 (0.71)
  Part 2: number analyzed (Participants) | 31 | 30
  Part 2 | 12.4 (1.75) | 12.8 (2.54)

5. Primary Outcome: Corneal Sensitivity
Description: The aesthesiometer will be used to perform corneal sensitivity to assess changes from baseline. Corneal Sensitivity Scale. Scale of 0-6
Time Frame: Part 1: 12 days time frame; Part 2: 35 days time frame
Population: Number analyzed comes from Part 2
Measure: Mean (Standard Deviation); unit: unit of measure "mm"
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
unit of measure "mm" | 59.8 (0.91) | 59.4 (1.74)

6. Primary Outcome: Undilated Fundoscopy
Description: Non-Contact undilated fundoscopy exam will be performed to assess changes from baseline; outcome measure is number of patients with no abnormalities
Time Frame: Part 2: 35 days time frame
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
Participants | 31 | 30

7. Primary Outcome: Vital Signs - Pulse
Description: Changes in vital signs is performed to assess changes from baseline
Time Frame: Part 1: 12 days time frame; Part 2: 35 days time frame
Population: Number analyzed comes from Part 1 and Part 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Active | Placebo
Number analyzed (Participants) | 37 | 32
beats per minute
  Part 1: number analyzed (Participants) | 6 | 2
  Part 1 | 64.3 (9.09) | 75.0 (4.24)
  Part 2: number analyzed (Participants) | 31 | 30
  Part 2 | 68.8 (10.55) | 70.5 (15.66)

8. Primary Outcome: Vital Signs - O2 Saturation
Description: Changes in vital signs is performed to assess changes from baseline
Time Frame: Part 1: 12 days time frame; Part 2: 35 days time frame
Population: Number analyzed comes from Part 1 and Part 2
Measure: Mean (Standard Deviation); unit: percentage of 02 saturation
Arm/Group | Active | Placebo
Number analyzed (Participants) | 37 | 32
percentage of 02 saturation
  Part 1: number analyzed (Participants) | 6 | 2
  Part 1 | 95.8 (1.94) | 97.0 (1.41)
  Part 2: number analyzed (Participants) | 31 | 30
  Part 2 | 96.3 (1.75) | 95.7 (1.66)

9. Primary Outcome: Vital Signs - Systolic Blood Pressure
Description: Changes in vital signs is performed to assess changes from baseline
Time Frame: Part 1: 12 days time frame; Part 2: 35 days time frame
Population: Number analyzed comes from Part 1 and Part 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
mmHg
  Part 1: number analyzed (Participants) | 6 | 2
  Part 1 | 128.0 (29.32) | 148.5 (3.54)
  Part 2: number analyzed (Participants) | 30 | 30
  Part 2 | 120.9 (15.97) | 128.2 (17.10)

10. Primary Outcome: Vital Signs - Diastolic Blood Pressure
Description: Changes in vital signs is performed to assess changes from baseline
Time Frame: Part 1: 12 days time frame; Part 2: 35 days time frame
Population: Number analyzed comes from Part 1 and Part 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
mmHg
  Part 1: number analyzed (Participants) | 6 | 2
  Part 1 | 72.7 (8.69) | 89.5 (9.19)
  Part 2 | 71.2 (9.53) | 72.0 (9.39)

11. Secondary Outcome: Ocular Discomfort
Description: Ocular discomfort Scale severity assessment (0-4 scale where 0 = none and 4 = constant)
Time Frame: Part 2: 35 days time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
score on a scale | 3.5 (0.78) | 3.9 (0.31)
Statistical Analysis 1: Comparison: Active vs Placebo; Change from Baseline. ANCOVA model includes baseline scores as a covariate; Test type: Superiority; p = 0.02, ANCOVA; Mean Difference (Net) = -0.3, 90% CI 2-sided [-0.7 to 0]

12. Secondary Outcome: Dry Eye Symptoms
Description: Dry eye syndrome symptom assessment Scale (grittiness) (0-5 scale where 0 = none and 5 = worst)
Time Frame: Part 2: 35 days time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
score on a scale | 1.7 (1.42) | 2.8 (1.38)
Statistical Analysis 1: Comparison: Active vs Placebo; Change form baseline. ANCOVA model includes baseline score as a covariate; Test type: Superiority; p = 0.0001, ANCOVA; Mean Difference (Net) = -1.0, 90% CI 2-sided [-1.4 to 0.5]

13. Secondary Outcome: Dry Eye Signs
Description: Dry eye syndrome staining Score assessments (total lissamine green staining score, 0-20 where 0 = no staining)
Time Frame: Part 2: 35 days time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
score on a scale | 5.88 (2.37) | 6.60 (2.55)
Statistical Analysis 1: Comparison: Active vs Placebo; Change from baseline. ANCOVA model includes baseline score as a covariate; Test type: Superiority; p = 0.03, ANCOVA; Mean Difference (Net) = -1.42, 90% CI 2-sided [-2.36 to -0.47]

14. Secondary Outcome: Tear Film Break up Time
Description: Tear film break up time measured (in seconds) after instillation of sodium fluorescein solution
Time Frame: Part 2: 35 days time frame
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
Seconds | 1.629 (0.85) | 1.480 (0.39)
Statistical Analysis 1: Comparison: Active vs Placebo; Change from Baseline; ANCOVA model includes baseline score as a covariate; Test type: Superiority; p = 0.39, ANCOVA; Mean Difference (Net) = 0.199, 90% CI 2-sided [-0.177 to 0.575]

15. Secondary Outcome: Schirmer's Test
Description: Measurement of Schirmer test strips (mm length of moistened area after 5 minutes)
Time Frame: Part 2: 35 days time frame
Measure: Mean (Standard Deviation); unit: mm in 5 minutes
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
mm in 5 minutes | 6.2 (4.19) | 6.7 (4.94)
Statistical Analysis 1: Comparison: Active vs Placebo; Change from baseline. ANCOVA model includes baseline score as a covariate; Test type: Superiority; p = 0.97, ANCOVA; Mean Difference (Net) = 0.2, 90% CI 2-sided [-1.7 to 2.0]

16. Secondary Outcome: Daily Symptom Assessment
Description: Daily symptom assessment using diary cards - outcome for worst symptom, ie symptom with highest severity score at baseline for each patient; calculated using the daily average between visit 3b to visit 4b Ora Calibra Ocular Discomfort & 4-Symptom Questionnaire (0-5 scale where 0 = none and 5 = worst)
Time Frame: Assessed daily between visit 3b (day 27) to visit 4b (day 35)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 31 | 30
score on a scale | 2.33 (0.832) | 2.69 (0.648)
Statistical Analysis 1: Comparison: Active vs Placebo; Change from baseline. ANCOVA model includes baseline score as a covariate; Test type: Superiority; p = 0.06, ANCOVA; Mean Difference (Net) = -0.23, 90% CI 2-sided [-0.48 to 0.03]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32
Other Adverse Events (participants affected / at risk) | 6/37 | 4/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=37) | Placebo (N=32)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1)
Eye Discharge (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Ocular itching (Eye disorders) | 1 (1) | 0 (0)
Instillation site pain (General disorders) | 1 (1) | 2 (2)
Instillation site discomfort (General disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Common cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03088605/Prot_002.pdf
  • Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT03088605/SAP_001.pdf